CLINICAL TRIAL: NCT02507713
Title: Ultrasound Markers for the Diagnosis, Disease Progression and Prognosis of Amyotrophic Lateral Sclerosis
Brief Title: Quantitative Neuromuscular Ultrasonography in Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALS
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jacinto Martínez-Payá, Professor of Human Anatomy and Biomedical Imaging, Universidad Católica San Antonio de Murcia
Other Study IDs: PMAFI10/14
Record Dates: First submitted 2015-07-20; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Ultrasonography; Motor neurons; Neuromuscular diseases; Fasciculation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Fasciculation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a progressive and fatal neurological disease. Nonspecific symptoms lead to a delay in the diagnosis, only confirmed by the electrophysiologic study.

Objectives.

1. To establish the diagnostic value of ultrasonography in ALS.
2. To evaluate the rate of muscle and nerve degeneration by ultrasonography in patients with ALS.
3. To check the relationship between ultrasound, clinical variables and functional tests in patients with ALS.

Methods. A longitudinal observational study in a consecutive sample of patients diagnosed with ALS will be realized. All the patients will be examined 3 times during 6 months and capabilities associated with ALS and muscle strength will be assessed. Bilateral and cross sectional ultrasonography of several muscles and also median and tibial nerves will be performed. All the images will be processed and analyzed for obtaining morphometric variables (muscle thickness and nerve area) and textural ones (echogenic variation, entropy, homogeneity, textural contrast and correlation). Frequency of twitches will be also recorded. After longitudinal study, a survival study will be performed in relation to functional and sonographic variables.

ELIGIBILITY:
Inclusion Criteria:

* Definite ALS.

Exclusion Criteria:

* Primary Lateral Sclerosis (PLS)
* Other forms of motor neuron disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with Amyotrophic Lateral Sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Measuring muscle thickness. | 6 months
  This measurement is carried out in the biceps brachialis, forearm flexors, quadriceps and tibialis anterior, which will be compared between patient with ALS and control group.

SECONDARY OUTCOMES:
Measurement muscle strength. | 6 months
  Graded on the medical research council scale
Measurement ALS Functional Rating Scale (ALSFRS-r) scale. | 6 months
  Recorded as the global score
Measurement muscle fasciculations. | 6 months
  Each muscle will be screened during 10 s.
Measuring muscle echointensity. | 6 months
  It will be measured using the Image J (v.1.48) software in the biceps brachialis, forearm flexors, quadriceps and tibialis anterior, which will be compared between patient with ALS and control group.
Measuring nerve area. | 6 months
  This measurement is carried out in the median and tibialis posterior nerves, which will be compared between patient with ALS and control group.

CONTACTS AND LOCATIONS:
Overall Officials: María E del Baño-Aledo, PhD, Principal Investigator — Human Anatomy Department. Universidad Católica San Antonio, Campus de los Jerónimos 138. 30107 Guadalupe, Murcia, Spain
Locations (1):
- Universidad Católica San Antonio de Murcia, Guadalupe, Murcia, Spain

REFERENCES:
- [Background] Cartwright MS, Walker FO, Griffin LP, Caress JB. Peripheral nerve and muscle ultrasound in amyotrophic lateral sclerosis. Muscle Nerve. 2011 Sep;44(3):346-51. doi: 10.1002/mus.22035. Epub 2011 Aug 3. PMID 21815172
- [Background] Schreiber S, Abdulla S, Debska-Vielhaber G, Machts J, Dannhardt-Stieger V, Feistner H, Oldag A, Goertler M, Petri S, Kollewe K, Kropf S, Schreiber F, Heinze HJ, Dengler R, Nestor PJ, Vielhaber S. Peripheral nerve ultrasound in amyotrophic lateral sclerosis phenotypes. Muscle Nerve. 2015 May;51(5):669-75. doi: 10.1002/mus.24431. Epub 2015 Mar 14. PMID 25155020
- [Background] Arts IM, Pillen S, Schelhaas HJ, Overeem S, Zwarts MJ. Normal values for quantitative muscle ultrasonography in adults. Muscle Nerve. 2010 Jan;41(1):32-41. doi: 10.1002/mus.21458. PMID 19722256
- [Result] Mayans D, Cartwright MS, Walker FO. Neuromuscular ultrasonography: quantifying muscle and nerve measurements. Phys Med Rehabil Clin N Am. 2012 Feb;23(1):133-48, xii. doi: 10.1016/j.pmr.2011.11.009. Epub 2011 Dec 9. PMID 22239880
- [Result] Arts IMP, Overeem S, Pillen S, Jurgen Schelhaas H, Zwarts MJ. Muscle changes in amyotrophic lateral sclerosis: a longitudinal ultrasonography study. Clin Neurophysiol. 2011 Mar;122(3):623-628. doi: 10.1016/j.clinph.2010.07.023. PMID 20810308
- [Result] Arts IM, Overeem S, Pillen S, Kleine BU, Boekestein WA, Zwarts MJ, Jurgen Schelhaas H. Muscle ultrasonography: a diagnostic tool for amyotrophic lateral sclerosis. Clin Neurophysiol. 2012 Aug;123(8):1662-7. doi: 10.1016/j.clinph.2011.11.262. Epub 2012 Jan 13. PMID 22244867
- [Result] Arts IM, Overeem S, Pillen S, Schelhaas HJ, Zwarts MJ. Muscle ultrasonography to predict survival in amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 2011 May;82(5):552-4. doi: 10.1136/jnnp.2009.200519. Epub 2010 Apr 14. PMID 20392981
- [Result] Pillen S, Arts IM, Zwarts MJ. Muscle ultrasound in neuromuscular disorders. Muscle Nerve. 2008 Jun;37(6):679-93. doi: 10.1002/mus.21015. PMID 18506712
- [Result] Arts IM, van Rooij FG, Overeem S, Pillen S, Janssen HM, Schelhaas HJ, Zwarts MJ. Quantitative muscle ultrasonography in amyotrophic lateral sclerosis. Ultrasound Med Biol. 2008 Mar;34(3):354-61. doi: 10.1016/j.ultrasmedbio.2007.08.013. Epub 2007 Oct 26. PMID 17964067
- [Result] Gdynia HJ, Muller HP, Ludolph AC, Koninger H, Huber R. Quantitative muscle ultrasound in neuromuscular disorders using the parameters 'intensity', 'entropy', and 'fractal dimension'. Eur J Neurol. 2009 Oct;16(10):1151-8. doi: 10.1111/j.1468-1331.2009.02663.x. Epub 2009 May 22. PMID 19486136